CLINICAL TRIAL: NCT02713360
Title: Screening and Intervention Reducing Anxiety in Patients With Implanted Cardioverter Defibrillator (ICD) - Screen-ICD
Brief Title: Screening and Intervention Reducing Anxiety in Patients With Implanted Cardioverter Defibrillator (ICD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Selina Kikkenborg Berg, Senior reseacher, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Screen-ICD
Record Dates: First submitted 2016-03-09; First posted 2016-03-18 (Estimated); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: ICD; Cognitive Therapy; Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive therapy (Experimental): The intervention consists of 3 steps. 1: Consultation with a nurse that aims of identifying what the anxiety consist of and how the patient experiences his or her life situation with an ICD. A plan is made to structure the treatment. 2: Participation in an individualized intervention based on anxiety type specific protocols. 3. The intervention is considered finalized if the patient has a HADS-A score under 8 two times in a row. The intervention group will receive usual care as well.
  Interventions: Behavioral: Cognitive Therapy
- Usual care (No Intervention): The control group will receive usual care which consists of control of ICD, disease control and treatment, and at one of the sites an offer of a group information meeting where experiences and events with ICD are discussed. The meeting takes place at Rigshospitalet every other month.

INTERVENTIONS:
Behavioral: Cognitive Therapy
  Arms: Cognitive therapy

SUMMARY:
The hypothesis is that there is a significant difference in anxiety scores between intervention and usual care group after intervention.

The aim of this randomised trial is (I) to determine the type of anxiety in ICD patients and (ii) to investigate the effect of screening followed by randomisation to intervention with consultations based on cognitive therapeutic principals to reduce anxiety in patients with ICD or usual care.

DETAILED DESCRIPTION:
Screen-ICD is an investigator-initiated randomised clinical superiority trial with blinded outcome assessment, including two university hospitals, with 1:1 randomisation to cognitive therapy plus usual care or usual care alone.

The intervention: all patients receive usual care. Patients in the intervention group will receive an intervention based on cognitive behavioral therapy. The intervention consists of three steps: 1. The intervention begins with a consultation with a nurse aiming at uncovering anxiety using the Hamilton anxiety scale and exploring how life with an ICD is perceived, 2. Based on the pre-specified protocols for each type of anxiety, cognitive therapy is provided and 3. After each session participants are asked to fill out the HADS questionnaire. When the patient scores below the cut-off value two times in a row, sessions will end. Each patient can have a maximum of 15 sessions.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years
* Have had ICD implantation
* Speaks and understands Danish
* Scores 8 or more in the HADS-A questionnaire
* Gives written informed consent

Exclusion Criteria:

* Scores 11 or more in the HADS-D questionnaire and the depression score exceeds the anxiety score.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
Primary outcome is anxiety measured by HADS. | 16 weeks
  HADS is a 14 item questionnaire that assesses anxiety and depression level in medical ill persons who are not admitted in psychiatric wards.
  Scores of 0 to 7 for either subscale are regarded as normal and scores of 8 to 10 suggest the presence of a mood disorder. Scores of 11 and above suggest probable presence of a mood disorder.

SECONDARY OUTCOMES:
Anxiety measured by HADS. | 12 months
  HADS is a 14 item questionnaire that assesses anxiety and depression level in medical ill persons who are not admitted in psychiatric wards.
  Scores of 0 to 7 for either subscale are regarded as normal and scores of 8 to 10 suggest the presence of a mood disorder. Scores of 11 and above suggest probable presence of a mood disorder.
Becks Anxiety Inventory (BAI) | 16 weeks and 12 months
  Becks Anxiety Inventory is a brief self-reported measure of anxiety with a focus on somatic symptoms of anxiety and was developed as a measure to discriminate between anxiety and depression. Respondents indicated how much each symptom has bothered them during the past week on a 4-point Likert scale ranging from 0 (not at all) to 3 (severely). The BAI score ranges from 0-63.
Hamilton Anxiety Scale (HAM-A) | 16 weeks and 12 months
  Hamilton Anxiety Scale is a clinical interview rating scale of the psychic (mental agitation and psychological distress) and somatic (physical complaints related to anxiety) aspects of anxiety. The scale consists of 14 clinical symptoms that are rated on a 5-point Likert scale ranging from 0 (not present) to 4 (very severe).
HeartQoL | 16 weeks and 12 months
  The questionnaire measures health-related quality of life in patients with ischemic heart disease, specifically angina, myocardial infarction or ischemic heart failure. The questionnaire consists of 14 items and provides two subscales; a 10-item physical subscale and a 4-item emotional subscale which are scored from 0 to 3.

OTHER OUTCOMES:
ICD Shock | 16 weeks and 12 months
  The number of ICD shocks will be evaluated within the 16 weeks and the data will be aggregated from the Danish Pacemaker & ICD Register.
Time to first schock | 16 weeks and 12 months
  Time to first schock will be measured within the 16 weeks in number of days and the data will be aggregated from the Danish Pacemaker & ICD Register.
Anti tachycardia pacing (ATP) | 16 weeks and 12 months
  The number of ATP will be evaluated within the 16 weeks and the data will be aggregated from the Danish Pacemaker & ICD Register.
Sleep quality | 16 weeks and 12 months
  Patients' own evaluation of sleep quality at 16 weeks and 12 months.
Physical activity | 16 weeks and 12 months
  Patients' own evaluation of physical activity at 16 weeks and 12 months.
Alcohol | 16 weeks and 12 months
  Number of alcohol units per week.
Smoking | 16 weeks and 12 months
  Number of cigarettes per day.
Weight | 16 weeks and 12 months
  Weight in kilogram.

CONTACTS AND LOCATIONS:
Overall Officials: Selina K. Berg, PhD., Principal Investigator — Rigshospitalet, Denmark
Locations (2):
- Denmark (2):
  - Rigshospitalet, Copenhagen
  - Herlev and Gentofte Hospital, Hellerup

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Berg SK, Herning M, Svendsen JH, Christensen AV, Thygesen LC. The Screen-ICD trial. Screening for anxiety and cognitive therapy intervention for patients with implanted cardioverter defibrillator (ICD): a randomised controlled trial protocol. BMJ Open. 2016 Oct 21;6(10):e013186. doi: 10.1136/bmjopen-2016-013186. PMID 27798030